CLINICAL TRIAL: NCT04808206
Title: A Multicentric Prospective Registry of Laparoscopic Bariatric Surgery Using Stapling Devices: Observation of Safety and Clinical Efficacy
Brief Title: A Registry of Laparoscopic Bariatric Surgery Using Stapling Devices: Observation of Safety and Clinical Efficacy
Acronym: STAP-JOLI
Status: Active, not recruiting | Type: Observational
Sponsor: Duomed (Industry)
Responsible Party: Sponsor
Other Study IDs: DM-PRO-ST2021
Record Dates: First submitted 2021-03-11; First posted 2021-03-22 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Roux-en-Y Gastric Bypass; Gastrostomy; Nissen Sleeve
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obese patients eligible for laparoscopic bariatric surgery
  Interventions: Device: easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical)

INTERVENTIONS:
Device: easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical) — Investigational device: easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical). Device for the creation of anastomoses during laparoscopic bariatric surgery manufactured by Ezisurg Medical.

SUMMARY:
The purpose of this observational registry is to evaluate the safety and the clinical efficacy of laparoscopic bariatric surgery using stapling devices (easyEndoTM Universal Linear Cutting Stapler and reloads from Ezisurg Medical). The goal of the study will be achieved by reporting peri- and postoperative complications and the clinical outcome after surgery in a prospectively maintained database.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age at registry entry
* Patient and investigator signed and dated the informed consent form prior to the index-procedure.
* Patient has a BMI ≥ 35 kg/m2, with one or more related co-morbidities.
* Patient has a BMI ≥ 40 kg/m2.
* Patient is eligible for laparoscopic bariatric surgery.

Exclusion Criteria:

* Patient is unable/unwilling to provide informed consent.
* Patient has a history of bariatric surgery.
* Patient is unable to comply with the registry protocol or the proposed follow-up visits.
* Patient has a contra-indication for laparoscopic bariatric surgery.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Obese patients eligible for laparoscopic bariatric surgery. This registry will collect data from 250 laparoscopic bariatric procedures in which anastomoses are created with the easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of laparoscopic bariatric surgery using stapling devices (easyEndoTM Universal Linear Cutting Stapler and reloads - Ezisurg Medical) | At index procedure
  Number of conversions, number of re-interventions and number of participants with (serious) adverse events ≥ grade II Clavien-Dindo.
Safety of laparoscopic bariatric surgery using stapling devices (easyEndoTM Universal Linear Cutting Stapler and reloads - Ezisurg Medical) | At discharge up to 1 week
  Number of re-interventions and number of participants with (serious) adverse events ≥ grade II Clavien-Dindo.
Safety of laparoscopic bariatric surgery using stapling devices (easyEndoTM Universal Linear Cutting Stapler and reloads - Ezisurg Medical) | Follow-up 1: 1 month after the procedure
  Number of re-interventions and number of participants with (serious) adverse events ≥ grade II Clavien-Dindo.
Safety of laparoscopic bariatric surgery using stapling devices (easyEndoTM Universal Linear Cutting Stapler and reloads - Ezisurg Medical) | Follow-up 2: 6 months after the procedure
  Number of re-interventions and number of participants with (serious) adverse events ≥ grade II Clavien-Dindo.
Safety of laparoscopic bariatric surgery using stapling devices (easyEndoTM Universal Linear Cutting Stapler and reloads - Ezisurg Medical) | Follow-up 3: 12 months after the procedure
  Number of re-interventions and number of participants with (serious) adverse events ≥ grade II Clavien-Dindo.
Safety of laparoscopic bariatric surgery using stapling devices (easyEndoTM Universal Linear Cutting Stapler and reloads - Ezisurg Medical) | Follow-up 4: 24 months after the procedure
  Number of re-interventions and number of participants with (serious) adverse events ≥ grade II Clavien-Dindo.

SECONDARY OUTCOMES:
Device performance | At index procedure
  Number of procedures with technical success
Device performance | At index procedure
  Scoring of: easy of intra-abdominal device positioning, grasping/climbing force, sharpness of the blades, staple-line formation, device stability, device maneuverability, device consistency and reliability, ergonomic design, hemostasis. Each of the aforementioned items receives a score from 0 to 4, with 0 indicating that the user is very unsatisfied and 4 indicating that the user is very satisfied.
Clinical efficacy - weight loss | Follow-up 1: 1 month after the procedure
  Weight loss
Clinical efficacy - weight loss | Follow-up 2: 6 months after the procedure
  Weight loss
Clinical efficacy - weight loss | Follow-up 3: 12 months after the procedure
  Weight loss
Clinical efficacy - weight loss | Follow-up 4: 24 months after the procedure
  Weight loss
Number of participants with a post-operative change of cormorbidities | Follow-up 3: 12 months after the procedure
  Comorbidities (diabetes mellitus, peripheral arterial disease, coronary arterial disease, sleep disordered breathing, hypertension, dyslipidemia, hypercholesterolemia, hypertriglyceridemia, asthma, congestive heart failure, degenerative joint disease, gastroesophageal reflux, chronic obstructive pulmonary disease, use of immunosuppressants) 12 months after the surgical procedure as compared to the patients' comorbidities at baseline.
Number of participants with a post-operative change of cormorbidities | Follow-up 4: 24 months after the procedure
  Comorbidities (diabetes mellitus, peripheral arterial disease, coronary arterial disease, sleep disordered breathing, hypertension, dyslipidemia, hypercholesterolemia, hypertriglyceridemia, asthma, congestive heart failure, degenerative joint disease, gastroesophageal reflux, chronic obstructive pulmonary disease, use of immunosuppressants) 24 months after the surgical procedure as compared to the patients' comorbidities at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Lobue, MD, Principal Investigator — Hôpital de Nivelles (groupe Jolimont), Haine-Saint-Paul, Belgium
Locations (3):
- Belgium (3):
  - Ziekenhuis Oost-Limburg, campus St.-Jan, Genk
  - Hôpital de Nivelles, groupe Jolimont, Haine-Saint-Paul
  - Ziekenhuis Maas en Kempen, Maaseik

IPD SHARING:
Plan to Share IPD: No